CLINICAL TRIAL: NCT03970720
Title: Restoration of Hypoglycemia Awareness With Metoclopramide
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Simon Fisher (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Simon Fisher, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00118549; 1R01DK118082-01A1 (NIH)
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hypoglycemia Unawareness
Keywords: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- T1DM - Unaware: Metoclopramide (Experimental): T1DM participants with hypoglycemia unawareness determined by a hypoglycemic clamp study will receive 10 mg metoclopramide four times a day during the four-week intervention period.
  Interventions: Drug: Metoclopramide
- T1DM - Unaware: Placebo (Placebo Comparator): T1DM participants with hypoglycemia unawareness determined by a hypoglycemic clamp study will receive 10 mg matching placebo capsules four times a day during the four-week intervention period.
  Interventions: Drug: Placebo
- T1DM - Aware: Placebo (Placebo Comparator): T1DM participants with hypoglycemia awareness determined by a hypoglycemic clamp study will receive 10 mg matching placebo capsules four times a day during the four-week intervention period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoclopramide — 10 mg metoclopramide four times a day
  Arms: T1DM - Unaware: Metoclopramide
Drug: Placebo — 10 mg matching placebo capsules four times a day
  Arms: T1DM - Aware: Placebo; T1DM - Unaware: Placebo

SUMMARY:
Metoclopramide is a drug approved by the FDA for gastroesophageal reflux and to relieve symptoms in adults with acute and recurrent diabetic gastroparesis. The objective of this study is to determine whether metoclopramide can improve hypoglycemia awareness and decrease the incidence of hypoglycemia in type 1 diabetes patients with hypoglycemia unawareness.

DETAILED DESCRIPTION:
Hypoglycemia is the most prevalent clinical complication in the daily management of diabetes and is the major obstacle to normalizing blood sugar. For people with Type 1 diabetes mellitus (T1DM), hypoglycemia associated autonomic failure (HAAF) increases the risk for severe hypoglycemia by a factor of 25 or more. A major component of HAAF is hypoglycemia unawareness (perhaps more accurately defined as impaired awareness of hypoglycemia), which involves in the loss/diminution of warning symptoms to hypoglycemia that would normally prompt a corrective behavioral response (e.g., eating food). Approximately 25-40% of people with T1DM report hypoglycemia unawareness. This value is most certainly an underestimation, as even people with diabetes who report having intact hypoglycemia, demonstrate impaired awareness of biochemically confirmed hypoglycemia. Although a major clinical problem for people with T1DM, it remains largely unknown what therapeutic agents could possibly be used to treat hypoglycemia unawareness.

With a goal of identifying existing biological compounds that could restore hypoglycemia awareness, laboratory drug screens were conducted using animal models. It was postulated that an ideal drug would markedly enhance the ability to sense hypoglycemia and trigger a potentially life-saving behavioral response (ie, alert the subject to increase food consumption). The vast majority of tested drugs did not restore hypoglycemia awareness (ie, did not restore blunted food intake response to hypoglycemia). Interestingly, of all the drugs tested, the dopamine antagonist metoclopramide consistently restored hypoglycemia awareness in several preclinical experiments. Additionally, metoclopramide also restored the impaired counterregulatory response to hypoglycemia in the animal model of HAAF.

This pilot phase II clinical trial (with placebo control) will be conducted to determine if FDA approved doses of Metaclopramdide can restore both, 1) hypoglycemia awareness, and 2) the sympathoadrenal response to hypoglycemia in patients with T1DM and hypoglycemia unawareness.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 1 Diabetes Mellitus
* Diabetes duration > 5 years
* Hemoglobin A1c ≤ 9%
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines

Exclusion Criteria:

* History of myocardial infarction, cardiac arrhythmia, congestive heart failure and coronary artery insufficiency
* History of stroke or brain disease
* History of genitourinary obstruction or urinary retention
* Advanced liver disease
* Active anemia with hemoglobin less than 11 g/dL
* Female in pregnancy or breastfeeding, or not able to practice effective contraception during the study period
* Uncontrolled mania or active major depressive disorder
* Previous allergic reaction or side effect to heparin use
* Contraindications to metoclopramide or conditions raising the risk for complication development to metoclopramide, such as hypersensitivity to metoclopramide, ongoing mechanical gastrointestinal obstruction, uncontrolled hypertension, pheochromocytoma, seizure disorders, Parkinson's disease, use of neuroleptics or antipsychotics within 6 months, use of benzodiazepines within the last month, active or recent (last 14 days) use of monoamine oxidase inhibitors or opioids, active alcohol or drug abuse, or other sedatives
* Participation in another study evaluating treatment for impaired awareness of hypoglycemia or hypoglycemia-associated autonomic failure in the last 30 days
* Current use of unblinded real-time Continuous Glucose Monitoring System
* Frequent need of acetaminophen administration

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Glucagon | 4 weeks
  Blood samples will be drawn from study participants during the initial hypoglycemic clamp study (Day 0) and during the second hypoglycemic clamp study (Day 28) following the 4-week intervention period. The average change in blood glucagon level will be compared between the study arms.
Change in Blood Epinephrine | 4 weeks
  Blood samples will be drawn from study participants during the initial hypoglycemic clamp study (Day 0) and during the second hypoglycemic clamp study (Day 28) following the 4-week intervention period. The average change in blood epinephrine level will be compared between the study arms.
Change in Blood Norepinephrine | 4 weeks
  Blood samples will be drawn from study participants during the initial hypoglycemic clamp study (Day 0) and during the second hypoglycemic clamp study (Day 28) following the 4-week intervention period. The average change in blood norepinephrine level will be compared between the study arms.
Change in Blood Cortisol | 4 weeks
  Blood samples will be drawn from study participants during the initial hypoglycemic clamp study (Day 0) and during the second hypoglycemic clamp study (Day 28) following the 4-week intervention period. The average change in blood cortisol level will be compared between the study arms.
Change in Blood Pancreatic Polypeptide | 4 weeks
  Blood samples will be drawn from study participants during the initial hypoglycemic clamp study (Day 0) and during the second hypoglycemic clamp study (Day 28) following the 4-week intervention period. The average change in blood pancreatic polypeptide level will be compared between the study arms.
Change in Hypoglycemia Symptom Recognition | 4 weeks
  Participant's self-reported symptoms of hypoglycemia will be obtained during the initial hypoglycemic clamp study (Day 0) and during the second hypoglycemic clamp study (Day 28) following the 4-week intervention period.

SECONDARY OUTCOMES:
Ratio of Self-Reported Hypoglycemic Episodes to Total Hypoglycemic Episodes | 6 weeks
  Participants will complete a report of all hypoglycemic events during the study surveillance periods. The average ratio of self-reported hypoglycemic episodes to total hypoglycemic episodes recorded by Continuous Glucose Monitoring (CGM) during these periods will be compared between the study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Fisher, MD, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cryer PE. Hypoglycemia-associated autonomic failure in diabetes. Handb Clin Neurol. 2013;117:295-307. doi: 10.1016/B978-0-444-53491-0.00023-7. PMID 24095133
- [Background] Cryer PE. Mechanisms of hypoglycemia-associated autonomic failure in diabetes. N Engl J Med. 2013 Jul 25;369(4):362-72. doi: 10.1056/NEJMra1215228. No abstract available. PMID 23883381
- [Background] Heller SR, Cryer PE. Reduced neuroendocrine and symptomatic responses to subsequent hypoglycemia after 1 episode of hypoglycemia in nondiabetic humans. Diabetes. 1991 Feb;40(2):223-6. doi: 10.2337/diab.40.2.223. PMID 1991573
- [Background] Schultes B, Schmid SM, Wilms B, Jauch-Chara K, Oltmanns KM, Hallschmid M. Lactate infusion during euglycemia but not hypoglycemia reduces subsequent food intake in healthy men. Appetite. 2012 Jun;58(3):818-21. doi: 10.1016/j.appet.2012.01.022. Epub 2012 Jan 28. PMID 22314041
- [Background] Schmid SM, Jauch-Chara K, Hallschmid M, Oltmanns KM, Born J, Schultes B. Short-term nocturnal hypoglycaemia increases morning food intake in healthy humans. Diabet Med. 2008 Feb;25(2):232-5. doi: 10.1111/j.1464-5491.2007.02347.x. PMID 18290864
- [Background] Dewan S, Gillett A, Mugarza JA, Dovey TM, Halford JC, Wilding JP. Effects of insulin-induced hypoglycaemia on energy intake and food choice at a subsequent test meal. Diabetes Metab Res Rev. 2004 Sep-Oct;20(5):405-10. doi: 10.1002/dmrr.471. PMID 15343587
- [Background] Towler DA, Havlin CE, Craft S, Cryer P. Mechanism of awareness of hypoglycemia. Perception of neurogenic (predominantly cholinergic) rather than neuroglycopenic symptoms. Diabetes. 1993 Dec;42(12):1791-8. doi: 10.2337/diab.42.12.1791. PMID 8243825
- [Background] Geddes J, Schopman JE, Zammitt NN, Frier BM. Prevalence of impaired awareness of hypoglycaemia in adults with Type 1 diabetes. Diabet Med. 2008 Apr;25(4):501-4. doi: 10.1111/j.1464-5491.2008.02413.x. PMID 18387080
- [Background] Kubiak T, Hermanns N, Schreckling HJ, Kulzer B, Haak T. Assessment of hypoglycaemia awareness using continuous glucose monitoring. Diabet Med. 2004 May;21(5):487-90. doi: 10.1111/j.1464-5491.2004.1136.x. PMID 15089796